CLINICAL TRIAL: NCT03715595
Title: The Treat-to-target Study of Rheumatoid Arthritis Based on Smart System of Disease Management(SSDM) : A Randomized Controlled Multicenter Trial
Brief Title: The Treat-to-target Study of RA Based on Smart System of Disease Management(SSDM)
Acronym: T2TRAonSSDM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Anhui Provincial Hospital (Other Government); The First Affiliated Hospital of Anhui Medical University (Other); Peking University International Hospital (Other); Xuanwu Hospital, Beijing (Other); Dongguan donghua hospital (Unknown); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Hebei General Hospital (Other); Bethune International Peace Hospital (Other); Central South University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Subei People's Hospital of Jiangsu Province (Other); The First Affiliated Hospital of BaoTou Medical College (Other); Linyi People's Hospital (Other); Shandong Provincial Hospital (Other Government); Mianyang Central Hospital (Other); Tianjin Medical University General Hospital (Other); The First People's Hospital of Yunnan (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Zhejiang Provincial People's Hospital (Other); First Hospital of China Medical University (Other); Xijing Hospital (Other); Tianjin First Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018PHB065-01
Record Dates: First submitted 2018-10-04; First posted 2018-10-23 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Rheumatoid Arthritis
Keywords: treat-to-target; smart system of disease management; drug use
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSDM group (Experimental): The patients in will use the SSDM at home every month for one year.
  Interventions: Other: SSDM group
- Control group (No Intervention): The patients will receive the conventional therapy for half a year. After half a year, all the patients will use the SSDM at home monthly for half a year.

INTERVENTIONS:
Other: SSDM group — The patients can perform self-evaluation, including DAS28, morning stiffness duration (MSD) and HAQ, and input medical records (including medication and laboratory test results) every month.
  Other Names: control group
  Arms: SSDM group

SUMMARY:
This study evaluate the Smart System of Disease Management（SSDM）to improve the treat-to-target(T2T) and the safety of drug in the treatment of rheumatoid(RA). All participants will be randomized in the SSDM group and the control group. The patients in the SSDM group will use the SSDM every month and the control group will receive the conventional therapy.

DETAILED DESCRIPTION:
Treat-to-Target (T2T), achieving a DAS28 score lower than 2.6 (remission, Rem) or below 3.2 (low disease activity, LDA), is the main management strategy recommended by ACR and EULAR. The Smart System of Disease Management (SSDM) is an interactive mobile disease management tool, including the doctors' and patients' application system. The patients can perform self-evaluation, including DAS28, morning stiffness duration (MSD) and HAQ, and input medical records (including medication and laboratory test results) through the mobile application. The data synchronizes to the mobiles of authorized rheumatologists through cloud data base and advices could be delivered.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Rheumatoid Arthritis.
2. Have a smartphone
3. Must be able to access disease activity by themselves

Exclusion Criteria:

1. Not able to access disease activity by themselves
2. Lacks the ability of self-management
3. Mental disorders or severe physical dysfunction
4. Extremely poor compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-05-29 (Estimated); Study Completion 2020-06-29 (Estimated)

PRIMARY OUTCOMES:
The rate of T2T between the two groups. | six month
  Self-reported data was reported at baseline and every month until the sixth month in the SSDM group and the patients only reported their disease at baseline and the sixth month in the control group.

SECONDARY OUTCOMES:
The rate of T2T between the two groups. | twelve month
  Self-reported data was reported every month until the twelve month in the two groups
The relapse rate between the two groups | Six month and twelve month
  Self-reported data was reported at baseline and every month until the sixth month in the SSDM group and the patients only reported their disease at baseline and the sixth month in the control group. After 6 months， all the patients will use the SSDM for 6 months.
The safety of drug use between the two groups | Six month and twelve month
  Self-reported data was reported at baseline and every month until the sixth month in the SSDM group and the patients only reported their disease at baseline and the sixth month in the control group. After 6 months， all the patients will use the SSDM for 6 months.
The compliance between the two groups | Six month and twelve month
  Self-reported data was reported at baseline and every month until the sixth month in the SSDM group and the patients only reported their disease at baseline and the sixth month in the control group. After 6 months， all the patients will use the SSDM for 6 months.
The HADS between the two groups | Six month and twelve month
  Self-reported data was reported at baseline and every month until the sixth month in the SSDM group and the patients only reported their disease at baseline and the sixth month in the control group. After 6 months， all the patients will use the SSDM for 6 months.
The SF-36 between the two groups | Six month and twelve month
  Self-reported data was reported at baseline and every month until the sixth month in the SSDM group and the patients only reported their disease at baseline and the sixth month in the control group. After 6 months， all the patients will use the SSDM for 6 months.
The medical economics between the two groups | Six month and twelve month
  Self-reported data was reported at baseline and every month until the sixth month in the SSDM group and the patients only reported their disease at baseline and the sixth month in the control group. After 6 months， all the patients will use the SSDM for 6 months.
The numbers of active intervention by doctors between the two groups | Six month and twelve month
  Self-reported data was reported at baseline and every month until the sixth month in the SSDM group and the patients only reported their disease at baseline and the sixth month in the control group. After 6 months， all the patients will use the SSDM for 6 months.
The effect of active intervention by doctors between the two groups | Six month and twelve month
  Self-reported data was reported at baseline and every month until the sixth month in the SSDM group and the patients only reported their disease at baseline and the sixth month in the control group. After 6 months， all the patients will use the SSDM for 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Chun Li, doctor, Study Director — Peking University People's Hospital
Locations (1):
- Chun Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barlow J, Turner A, Swaby L, Gilchrist M, Wright C, Doherty M. An 8-yr follow-up of arthritis self-management programme participants. Rheumatology (Oxford). 2009 Feb;48(2):128-33. doi: 10.1093/rheumatology/ken429. Epub 2008 Nov 26. PMID 19036778
- [Result] McBain H, Shipley M, Olaleye A, Moore S, Newman S. A patient-initiated DMARD self-monitoring service for people with rheumatoid or psoriatic arthritis on methotrexate: a randomised controlled trial. Ann Rheum Dis. 2016 Jul;75(7):1343-9. doi: 10.1136/annrheumdis-2015-207768. Epub 2015 Aug 19. PMID 26290587
- [Result] Dougados M, Soubrier M, Perrodeau E, Gossec L, Fayet F, Gilson M, Cerato MH, Pouplin S, Flipo RM, Chabrefy L, Mouterde G, Euller-Ziegler L, Schaeverbeke T, Fautrel B, Saraux A, Chary-Valckenaere I, Chales G, Dernis E, Richette P, Mariette X, Berenbaum F, Sibilia J, Ravaud P. Impact of a nurse-led programme on comorbidity management and impact of a patient self-assessment of disease activity on the management of rheumatoid arthritis: results of a prospective, multicentre, randomised, controlled trial (COMEDRA). Ann Rheum Dis. 2015 Sep;74(9):1725-33. doi: 10.1136/annrheumdis-2013-204733. Epub 2014 May 28. PMID 24872377
- [Result] Harrison BJ, Symmons DP, Brennan P, Barrett EM, Silman AJ. Natural remission in inflammatory polyarthritis: issues of definition and prediction. Br J Rheumatol. 1996 Nov;35(11):1096-100. doi: 10.1093/rheumatology/35.11.1096. PMID 8948295
- [Result] Krishna S, Boren SA, Balas EA. Healthcare via cell phones: a systematic review. Telemed J E Health. 2009 Apr;15(3):231-40. doi: 10.1089/tmj.2008.0099. PMID 19382860
- [Result] Marshall A, Medvedev O, Antonov A. Use of a smartphone for improved self-management of pulmonary rehabilitation. Int J Telemed Appl. 2008;2008:753064. doi: 10.1155/2008/753064. PMID 18615186
- [Result] Azevedo R, Bernardes M, Fonseca J, Lima A. Smartphone application for rheumatoid arthritis self-management: cross-sectional study revealed the usefulness, willingness to use and patients' needs. Rheumatol Int. 2015 Oct;35(10):1675-85. doi: 10.1007/s00296-015-3270-9. Epub 2015 Apr 24. PMID 25903352
- [Derived] Li C, Huang J, Wu H, Li F, Zhao Y, Zhang Z, Li S, Wei H, Zhang M, Sun H, Yang J, Li Q, Li X, Qi W, Wei W, Li Y, Li Z, Wang Y, Zhang F, Wu H, Shuai Z, Wu Z, Li Y, Jia S, Jia Y, Xiao F, Mu R, Li Z. Management of Rheumatoid Arthritis With a Digital Health Application: A Multicenter, Pragmatic Randomized Clinical Trial. JAMA Netw Open. 2023 Apr 3;6(4):e238343. doi: 10.1001/jamanetworkopen.2023.8343. PMID 37058302